CLINICAL TRIAL: NCT02940119
Title: Effects of Phototherapy With Different Sources of Light in Muscle Skeletal Chronic Pain Relief From Neck and Shoulders
Brief Title: Neck and Shoulder Pain Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 041016
Record Dates: First submitted 2016-10-04; First posted 2016-10-20 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Neck Pain; Shoulder Pain; Chronic Pain; Musculoskeletal Pain
MeSH Terms: conditions — Neck Pain; Shoulder Pain; Chronic Pain; Musculoskeletal Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Active PBMT (Active Comparator): The volunteers received active phototherapy in each session.
  Interventions: Device: Multi Radiance Medical®
- Placebo PBMT (Placebo Comparator): The volunteers received placebo phototherapy in each session.
  Interventions: Device: Multi Radiance Medical®

INTERVENTIONS:
Device: Multi Radiance Medical® — Volunteers received all procedures of the study with active or placebo phototherapy (PBMT) in 9 sites of the neck and shoulders, twice a week. The PBMT was applied in all sessions.
  Other Names: Photobiomodulation therapy

SUMMARY:
Pain in the neck and shoulders is a musculoskeletal disorder that affects a significant number of individuals.The aim of this study is to evaluate the effects of PBMT (with a device that combines low level laser therapy and light emitting diode therapy) in chronic pain relief of musculoskeletal origin in the neck and shoulders area.

DETAILED DESCRIPTION:
Randomized, placebo-controlled, double-blind clinical trial was carried out. Seventy-two patients with chronic pain in neck and shoulder were recruited and randomized into two groups (n = 36 each group), one group received active PBMT and another group received placebo PBMT (with a device with same appearance of the actual laser, including any visible light). Patients were treated at 9 different sites of 3 zones in the neck and shoulders area, twice a week during 3 consecutive weeks with a PBMT device manufactured by Multi Radiance Medical™ (Solon - OH, USA). Primary outcome was intensity of pain using the Visual Analog Pain Scale (VAS), secondary outcomes were range of motion (ROM) of the neck and shoulders and patient satisfaction with therapy employed.

Sample Size calculation: The success criterion was defined as a 30% or greater reduction in VAS from baseline to the final evaluation and overall efficacy of the PBMT/sMF therapy was considered successful if a minimal difference of 35% is found between the active and placebo group. It was anticipated that about 55% of subjects in the active group and about 20% of subjects in the placebo group would meet the individual success criteria and intended application of a two-tailored test with an alpha of 0.05 and power of 0.8.

A sample size of 33 eligible subjects per group was calculation31 and a subject loss-to-follow-up of 10% was anticipated to bring the sample size to 36 subjects in each group. To ensure statistically valid and representative data of the general population sampled, a total of 72 subjects were enrolled in this study and stratified by Fitzpatrick skin type as following: Lighter skinned individuals were into Fitzpatrick skin types I, II and III, while darker skinned individuals were into Fitzpatrick skin types IV, V and VI.

ELIGIBILITY:
Inclusion Criteria:

* presenting primary pain is located in the region of the neck (right side and/or left side and/or the back of the neck) and/or the shoulder (right side and/or left side);
* neck and/or shoulder pain is of benign musculoskeletal origin wherein the etiology is sprain strain and/or muscle spasms;
* neck/shoulder pain is episodic chronic, defined as having occurred and recurred over regular or irregular periods or intervals of time, persisting over at least the last 3 months;
* self-reported Degree of Pain rating on the 0-100 VAS pain scale for the neck-shoulder region is 50 or greater;
* subject is willing and able to maintain his or her current pre-study neck/shoulder pain management regimen of pain relief medication and/or treatment/therapy use throughout the course of study duration, whilst refraining from consuming other types of medication and/or prescription medication(s) and/or herbal supplements intended for the relief of pain and/or inflammation, including muscle relaxants, and/or partaking in other treatments/therapies including conventional therapies such as physical therapy, occupational therapy and hot or cold packs, as well as alternative therapies such as chiropractic care and acupuncture.

Exclusion Criteria:

* subject's presenting primary pain is located outside or in addition to the region of the neck (right side and/or left side and/or the back of the neck) and/or the shoulder (right side and/or left side);
* subject's neck and/or shoulder pain is of other than, or in addition to, benign musculoskeletal origin wherein the etiology is sprain strain and/or muscle spasms, and/or the etiology of the subject's neck/shoulder pain cannot be satisfactorily ruled out as one or more;
* neck/shoulder pain is acute, defined as having persisted over less than the last 3 months;
* neck/shoulder pain is not episodic, such that it has either been continually present without respite over the past 3 months and/or there has not been recurrent episodes within the past 3 months;
* self-reported Degree of Pain rating on the 0-100 VAS pain scale for the neck-shoulder region is less than 50;
* local corticosteroids and/or botulinum toxin (Botox®) injection for neck/shoulder pain relief within the prior 30 days;
* such as chiropractic care and acupuncture;
* current, active chronic pain disease: chronic fatigue syndrome, fibromyalgia, endometriosis, inflammatory bowel disease, interstitial cystitis diabetic neuropathic pain;
* cancer or treatment for cancer in the past 6 months, including tumors of the spinal cord, diabetes Type 1, significant heart conditions including coronary heart failure and implantable heart devices such as a pacemaker, active infection, wound or other external trauma to the areas to be treated with the laser, surgery to the neck and/or shoulder region in the past 12 months;
* medical, physical, or other contraindications for, or sensitivity to, light therapy;
* pregnant, breast feeding, or planning pregnancy prior to the end of study participation, serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years;
* developmental disability or cognitive impairment that in the opinion of the investigator would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements;
* involvement in litigation and/or receiving disability benefits related in any way to the parameters of the study;
* subject is less than 18 years of age;
* participation in a clinical study or other type of research in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pain assessment | one month
  Visual anagogic scale (VAS)

SECONDARY OUTCOMES:
Rage of Motion (ROM) | one month
  pre-defined assessment with a goniometer
Individualized pain management regimen | one month
  questionnaire about perception and what kind of phototherapy was performed (active or placebo). This assessment was answered by subjects, investigator that performed the assessments and investigator that performed phototherapy application.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Leal-Junior, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Laboratory of Phototherapy in Sports and Exercise, Universidade Nove de Julho (UNINOVE), São Paulo, São Paulo, Brazil